CLINICAL TRIAL: NCT00057330
Title: A Double-Blind, Randomized, Controlled Phase III Study to Assess the Prophylactic Efficacy and Safety of gD-Alum/MPL Vaccine in the Prevention of Genital Herpes Disease in Young Women Who Are HSV-1 and -2 Seronegative
Brief Title: HerpeVac Trial for Young Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208141/039; 208141/039 (Other: GSK)
Record Dates: First submitted 2003-03-31; First posted 2003-04-01 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2013-05

CONDITIONS: Herpes Simplex Infection
MeSH Terms: conditions — Herpes Simplex | interventions — Hepatitis A Vaccines; halofantrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Herpes Simplex Virus Group (Experimental): Females between, and including, 18 and 30 years of age at the time of first vaccination who received 3 doses of herpes simplex virus (HSV) vaccine intramuscularly in the non-dominant deltoid on a 0, 1, 6 month schedule.
  Interventions: Biological: HSV vaccine or SB208141, GSK Biologicals' glycoprotein D (gD)-Alum/3-deacylated form of Monophosphoryl Lipid A (MPL) candidate genital herpes vaccine
- Havrix Group (Experimental): Females between, and including, 18 and 30 years of age at the time of first vaccination who received 3 doses of the investigational formulation of Havrix vaccine intramuscularly in the non-dominant deltoid on a 0, 1, 6 month schedule.
  Interventions: Biological: Havrix™, GlaxoSmithKline (GSK) Biologicals' licensed Hepatitis A vaccine

INTERVENTIONS:
Biological: HSV vaccine or SB208141, GSK Biologicals' glycoprotein D (gD)-Alum/3-deacylated form of Monophosphoryl Lipid A (MPL) candidate genital herpes vaccine — the vaccine was administered intramuscularly in the non-dominant deltoid
  Arms: Herpes Simplex Virus Group
Biological: Havrix™, GlaxoSmithKline (GSK) Biologicals' licensed Hepatitis A vaccine — the vaccine was administered intramuscularly in the non-dominant deltoid
  Arms: Havrix Group

SUMMARY:
The primary purpose of this study is to see if a herpes vaccine may prevent genital herpes disease in women who are not infected. The study will enroll approximately 7550 healthy women. These women will be randomly assigned to 1 of 2 possible study groups: herpes vaccine (experimental group) or hepatitis A vaccine (control group). Participants will receive their assigned vaccine at 0, 1, and 6 months. Participants will have 9 scheduled study visits and additional unscheduled visits for an evaluation of herpes if it is suspected. Participants will be involved in study related procedures for up to 20 months.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, controlled Phase III trial to assess the prophylactic efficacy and safety of gD-Alum/MPL vaccine in the prevention of genital herpes disease in young women who are herpes simplex virus (HSV)-1 and -2 seronegative. The primary efficacy objective is to evaluate vaccine efficacy in the prevention of genital herpes disease caused by HSV-1 and/or HSV-2 between months 2 and 20 in healthy adult women who were initially HSV-1 and HSV-2 seronegative. The secondary efficacy objectives are to: evaluate vaccine efficacy in the prevention of genital herpes disease caused by HSV-1 and/or HSV-2 occurring between the months 7 and 20; evaluate vaccine efficacy in the prevention of HSV-2 infection between months 2 and 20; and to evaluate vaccine efficacy in the prevention of HSV-2 infection occurring between months 7 and 20. The study will enroll approximately 7,550 women, ages 18-30 years. Participants will be randomized to 1 of 2 possible study groups: candidate vaccine; or control vaccine (hepatitis A vaccine). The study duration for each subject will be approximately 20 months. Study procedures will include 9 scheduled study visits (including the screening visit) and additional unscheduled visits for evaluation of suspected herpes disease episodes. Three doses of vaccine or control will be administered intramuscularly in the non-dominant deltoid on a 0, 1, and 6 month schedule. Subjects will attend clinic visits at screening, months 2, 7, 12, 16, and 20. In subjects who present with suspected herpes disease between months 17 and 20, an additional visit to collect a serum sample will be scheduled 3 months after the evaluation for suspected genital herpes.

ELIGIBILITY:
Inclusion Criteria:

* A female between, and including, 18 and 30 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Seronegative for HSV-1 and HSV-2 by Western blot.
* Subject must be non-childbearing potential, i.e. either surgically sterilized or, if of child bearing potential, she must be using a highly effective method of birth control (e.g., intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant®; DepoProvera®; contraceptive skin patch or cervical ring) for 30 days prior to vaccination, have a negative urine pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
* A subject for whom the investigator believes can and will comply with the requirements of the protocol (e.g. completion of the memory aid/diary cards, return for follow-up visits, accessible by phone or pager, able to self-sample and not planning on moving from study area).

Exclusion Criteria:

* Pregnant or nursing female.
* Clinical signs or symptoms of current oro-labial, genital or non-genital HSV disease, such as swelling, papules, vesicles, pustules, ulcers, crusts, fissures, erythema, discharge, pain, burning, itching, tingling or dysuria.
* Previous vaccination against herpes.
* Previous administration of monophosphoryl lipid A (MPL) adjuvant (no vaccines currently licensed in the USA contain this).
* History of any confirmed oro-labial, genital or non-genital HSV disease or infection.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a non-study vaccine within 30 days of the first dose of the study vaccine with the following exceptions: Administration of routine Meningococcal, Hepatitis B, inactivated Influenza, and Diphtheria/Tetanus vaccine up to 8 days before the first dose of study vaccine is allowed.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines, e.g. aluminum, MPL, alum-MPL, 2-phenoxyethanol or neomycin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including, human immunodeficiency virus (HIV) infection.
* Acute or chronic, clinically significant (unresolved, requiring on-going medical management or medication, etc.) pulmonary, cardiovascular, hepatic or renal function abnormality, as determined by medical history or physical examination.
* Acute disease at the time of enrollment (defer vaccination until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever. Study vaccine can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness.
* Oral temperature greater than or equal to 99.5º F (greater than or equal to 37.5º C) / axillary temperature greater than or equal to 99.5º (greater than or equal to 37.5º C) / tympanic temperature on oral setting greater than or equal to 99.5º F (greater than or equal to 37.5º C).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. (For corticosteroids, this will mean prednisone or, equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled or topical steroids are allowed.)
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Recent history of chronic alcohol consumption (defined as more than 5 oz of ethanol [absolute alcohol] per day) and/or drug abuse.
* History of sexually transmitted infection within 30 days preceding the first dose of study vaccine.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8323 (Actual)
Dates: Start 2003-01-14; Primary Completion 2009-08-22 (Actual); Study Completion 2009-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (59):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Carson, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Satesboro, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Bloomington, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, College Park, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Grove City, Pennsylvania
  - GSK Investigational Site, Johnstown, Pennsylvania
  - GSK Investigational Site, Monongahela, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Kingston, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, La Crosse, Wisconsin
- Canada (8):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Beauport, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Derived] Belshe RB, Blevins TP, Yu Y, Nethington AE, Bellamy A, Bryant C, Morrison LA. Neutralizing Antibody Kinetics and Immune Protection Against Herpes Simplex Virus 1 Genital Disease in Vaccinated Women. J Infect Dis. 2023 Feb 14;227(4):522-527. doi: 10.1093/infdis/jiac067. PMID 35199165
- [Derived] Belshe RB, Heineman TC, Bernstein DI, Bellamy AR, Ewell M, van der Most R, Deal CD. Correlate of immune protection against HSV-1 genital disease in vaccinated women. J Infect Dis. 2014 Mar;209(6):828-36. doi: 10.1093/infdis/jit651. Epub 2013 Nov 27. PMID 24285844
- [Derived] Belshe RB, Leone PA, Bernstein DI, Wald A, Levin MJ, Stapleton JT, Gorfinkel I, Morrow RL, Ewell MG, Stokes-Riner A, Dubin G, Heineman TC, Schulte JM, Deal CD; Herpevac Trial for Women. Efficacy results of a trial of a herpes simplex vaccine. N Engl J Med. 2012 Jan 5;366(1):34-43. doi: 10.1056/NEJMoa1103151. PMID 22216840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8323 subjects were enrolled and vaccinated (4577 in the Herpes Simplex Virus Group and 3746 in the Havrix Group). Out of these, 7850 subjects were followed throughout the entire study, e. a. for safety and adverse event assessment (4488 in the Herpes Simplex Virus Group and 3662 in the Havrix Group).
Groups:
- Herpes Simplex Virus Group: Females between, and including, 18 and 30 years of age at the time of first vaccination who received 3 doses of herpes simplex virus vaccine (HSV) intramuscularly in the non-dominant deltoid on a 0, 1, 6 month schedule.
Period: Overall Study
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Started | 4577 | 3746
Completed | 3445 | 2826
Not Completed | 1132 | 920
Not completed — Adverse Event | 9 | 12
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 115 | 84
Not completed — Lost to Follow-up | 745 | 617
Not completed — Physician Decision | 1 | 0
Not completed — Other | 260 | 206

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Herpes Simplex Virus Group | Havrix Group | Total
Number analyzed (Participants) | 4577 | 3746 | 8323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.3 (3.30) | 22.3 (3.23) | 22.3 (3.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4577 | 3746 | 8323
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Newly Acquired Genital Herpes Disease, Caused by Either Herpes Simplex Virus (HSV)-1 or HSV-2
Description: Genital herpes disease was defined as signs (swelling, papules, vesicles, ulcers, crusts, fissures, erythema, or vaginal discharge) and/or symptoms (pain, burning, itching, tingling, dysuria) which developed on the skin or mucosa of the anogenital region and/or buttocks and laboratory confirmation of Herpes Simplex Virus (HSV)-1 or 2 infection (either concomitant positive HSV culture or HSV seroconversion within 6 months after onset of signs and/or symptoms). Seroconversion to HSV-1 and/or HSV-2 was defined as a positive HSV-1 and/or HSV-2 Western blot in a subject with a previously negative Western blot result for the corresponding HSV type.
Time Frame: Between Months 2 and 20
Population: The Per Protocol cohort for analysis of efficacy (Months 2-20) included all subjects who met inclusion/exclusion criteria, did not meet infection/disease, did not meet censoring criteria, had at least 1 efficacy assessment, received 2 doses of the vaccine within the permitted time interval, with known vaccine administration site and route.
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 3798 | 3076
Subjects | 35 | 35

2. Secondary Outcome: Number of Subjects With Newly Acquired Genital Herpes Disease, Caused by Either Herpes Simplex Virus (HSV)-1 or HSV-2
Description: as for outcome 1
Time Frame: Between Months 7 and 20
Population: The Per Protocol cohort for analysis of efficacy (Months 7-20) included all subjects who met inclusion/exclusion criteria, did not meet infection/disease, did not meet censoring criteria, had at least 1 efficacy assessment, received 3 doses of the vaccine within the permitted time interval, with known vaccine administration site and route.
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 3273 | 2622
Subjects | 18 | 22

3. Secondary Outcome: Number of Subjects With Newly Acquired Herpes Simplex Virus (HSV)-2 Infection Confirmed by Either Virus Culture or HSV-2 Seroconversion.
Description: The number of subjects with newly acquired HSV-2 infection confirmed by either virus culture or HSV-2 seroconversion was tabulated. Seroconversion to HSV-1 and/or HSV-2 was defined as a positive HSV-1 and/or HSV-2 Western blot in a subject with a previously negative Western blot result for the corresponding HSV type.
Time Frame: Between Months 2 and 20
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 3798 | 3076
Subjects | 62 | 46

4. Secondary Outcome: Number of Subjects With Newly Acquired Herpes Simplex Virus (HSV)-2 Infection Confirmed by Either Virus Culture or HSV-2 Seroconversion
Description: as for outcome 3
Time Frame: Between Months 7 and 20
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 3273 | 2622
Subjects | 40 | 35

5. Secondary Outcome: Concentrations for Anti-glycoprotein D (Anti-gD) Antibodies.
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA units per milliliter (EU/mL). The seroprotection cut-off of the assay was 40 EU/mL
Time Frame: At Months 0, 2, 6, 7, 12, 16 and 20
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects (meeting eligibility criteria, complying with protocol-defined procedures and not meeting either the infection or disease criteria on or prior to Month 7) for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 641 | 223
EU/mL
  Anti-gD GMCs at Month 0 | 21.52 [20.77 to 22.29] | 20.62 [19.94 to 21.32]
  Anti-gD GMCs at Month 2 | 3575 [3256 to 3925] | 21.39 [20.33 to 22.51]
  Anti-gD GMCs at Month 6 | 681.3 [622.1 to 746.2] | 21.58 [20.42 to 22.81]
  Anti-gD GMCs at Month 7 | 6809 [6344 to 7309] | 21.50 [20.36 to 22.71]
  Anti-gD GMCs at Month 12 | 1805 [1667 to 1955] | 21.14 [19.89 to 22.48]
  Anti-gD GMCs at Month 16 | 1025 [941.9 to 1115] | 20.10 [19.90 to 20.30]
  Anti-gD GMCs at Month 20 | 769.1 [704.1 to 840.0] | 20.60 [19.65 to 21.61]

6. Secondary Outcome: Titers for Anti-herpes Simplex Virus (Anti-HSV) Neutralizing Antibodies.
Description: Titers for Anti-HSV neutralizing antibodies are presented as Geometric Mean Titers (GMTs), and are expressed in Estimated Doses (ED), that is, the reciprocal of the dilution necessary to achieve neutralization. Antibody titers below the lowest level of quantification were not calculated .
Time Frame: At Months 0, 2, 6, 7, 12, 16 and 20
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ED
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 641 | 223
ED
  Anti-HSV GMTs at Month 0 | 2.09 [2.04 to 2.14] | 2.06 [2.00 to 2.12]
  Anti-HSV GMTs at Month 2 | 7.57 [6.86 to 8.34] | NA [NA to NA] — Antibody titers below the lowest level of quantification were not calculated.
  Anti-HSV GMTs at Month 6 | 2.42 [2.31 to 2.54] | NA [NA to NA] — Antibody titers below the lowest level of quantification were not calculated.
  Anti-HSV GMTs at Month 7 | 28.27 [26.59 to 30.06] | 2.10 [2.00 to 2.21]
  Anti-HSV GMTs at Month 12 | 8.40 [7.63 to 9.24] | 2.02 [1.99 to 2.05]
  Anti-HSV GMTs at Month 16 | 4.72 [4.32 to 5.16] | 2.03 [1.98 to 2.08]
  Anti-HSV GMTs at Month 20 | 3.65 [3.37 to 3.96] | 2.11 [2.01 to 2.22]

7. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling.
  Solicited general symptoms assessed were fatigue, headache, malaise and fever (defined as oral/axillary/tympanic temperature equal to or above 37.5 degrees Celsius).
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: The Intention To Treat cohort for the analysis of safety included all vaccinated subject for whom safety data were available.
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 4488 | 3662
Subjects
  Pain | 3902 | 2559
  Redness | 1621 | 702
  Swelling | 1371 | 438
  Fatigue | 2031 | 1503
  Headache | 1885 | 1456
  Malaise | 1459 | 1003
  Fever | 400 | 260

8. Secondary Outcome: Number of Subjects Reporting Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling.
  Grade 3 pain = pain that prevented normal activities.
  Grade 3 redness/swelling = redness/swelling above 30 mm and persisting for more than 24 hours
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 4488 | 3662
Subjects
  Grade 3 Pain | 307 | 67
  Grade 3 Redness | 40 | 2
  Grade 3 Swelling | 82 | 4

9. Secondary Outcome: Number of Subjects Reporting Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, headache, malaise and fever (oral/axillary/tympanic).
  Grade 3 headache, fatigue, malaise = symptom that prevented normal activities.
  Grade 3 fever = temperature above 39.0 degrees Celsius.
  Related = symptom assessed by the investigator as causally related to the vaccination
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 4488 | 3662
Subjects
  Grade 3 Fatigue | 225 | 146
  Fatigue related to vaccination | 1776 | 1286
  Grade 3 Headache | 175 | 126
  Headache related to vaccination | 1523 | 1171
  Grade 3 Malaise | 199 | 121
  Malaise related to vaccination | 1225 | 816
  Grade 3 Fever | 17 | 7
  Fever related to vaccination | 295 | 198

10. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs have been tabulated for a 31-day period. An unsolicited AE was any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31 days after vaccination
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 4488 | 3662
Subjects | 2154 | 1677

11. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCDs), Medically Significant Conditions (MSCs) and Serious Adverse Events (SAEs)
Description: NOCDs included adverse events (AEs) as autoimmune disorders, asthma, type I diabetes, allergies. MSCs included AEs prompting emergency room or physician visits unrelated to common diseases or routine visits for physical examination or vaccination, or SAEs unrelated to common diseases. SAEs included medical occurrences either life-threatening, requiring hospitalization, or resulting in death, disability/incapacity or congenital anomaly/birth defect in a subject's offspring. Common diseases included upper respiratory infections (URIs), sinusitis, pharyngitis, gastroenteritis, urinary tract infection, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury. The following were not reported if not considered as SAEs and occurring more than 30 days post vaccination: URIs, sinusitis, pharyngitis, gastroenteritis, injury, or visits for routine physical examination or vaccination. AEs are described, using Medical Dictionary for Regulatory Activities' preferred terms.
Time Frame: Throughout the study (From Month 0 up to Month 20)
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 4488 | 3662
Subjects
  NOCDs/MSCs/SAEs | 208 | 182
  Asthma | 14 | 16
  Abortion spontaneous | 24 | 13
  Hypothyroidism | 7 | 11
  Appendicitis | 5 | 9
  Hypoesthesia | 3 | 6
  Suicide attempt | 0 | 7
  Ovarian cyst | 0 | 4
  Meningitis viral | 0 | 3
  Dehydration | 0 | 3
  Depression | 6 | 3
  Suicidal ideation | 0 | 3
  Nephrolithaiasis | 0 | 3
  Premature labor | 0 | 4
  Pyelonephritis | 0 | 3
  Pyrexia | 3 | 0
  Pneumonia | 3 | 0
  Road traffic accident | 4 | 0
  Skin laceration | 3 | 0
  Abortion missed | 4 | 0
  Abortion spontaneous complete | 4 | 0
  Bipolar disorder | 5 | 0
  Depression suicidal | 3 | 0
  Crohn's disease | 0 | 3
  Hyperemesis gravidarum | 0 | 3
  Hyperthyroidism | 0 | 3

12. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in a subject's offspring.
Time Frame: Throughout the study (From Month 0 up to Month 20)
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Number analyzed (Participants) | 4488 | 3662
Subjects | 171 | 132

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Day 0-6) follow-up period after vaccination. Unsolicited adverse events: during the 31 days following vaccination period. Serious adverse events: from Month 0 up to Month 20
Description: Related SAEs were reported for 6 and 5 subjects in the Herpes Simplex Virus and Havrix groups, respectively. 1 fatal SAE was reported for 1 subject in the Herpes Simplex Virus Group, and assessed by the investigator as not related to vaccination.
Arm/Group | Herpes Simplex Virus Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 171/4488 | 132/3662
Other Adverse Events (participants affected / at risk) | 4133/4488 | 3061/3662
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herpes Simplex Virus Group (N=4488) | Havrix Group (N=3662)
Abortion spontaneous (Nervous system disorders) | 24 | 13 — This SAE was assessed the investigators as related to vaccination for 2 and one subjects in the Herpes Simplex Virus and Havrix groups, respectively.
Appendicitis (Infections and infestations) | 5 | 9
Depression (Psychiatric disorders) | 6 | 3
Suicide attempt (Psychiatric disorders) | 2 | 6
Bipolar disorder (Psychiatric disorders) | 4 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 2
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 4 | 1
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 4 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 3
Ovarian cyst (Reproductive system and breast disorders) | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Infectious mononucleosis (Infections and infestations) | 2 | 2 — This SAE was assessed the investigators as related to study vaccination for one subject in the Havrix Group.
Meningitis viral (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 3 | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 3
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 2 — This SAE was assessed the investigators as related to study vaccination for one subject in the Herpes Simplex Virus Group.
Anaphylactic reaction (Immune system disorders) | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Bipolar i disorder (Psychiatric disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Depression suicidal (Psychiatric disorders) | 3 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Migraine (Nervous system disorders) | 1 | 2
Ovarian cyst ruptured (Reproductive system and breast disorders) | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 3
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Chest pain (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0
Convulsion (Nervous system disorders) | 0 | 2
Endometriosis (Reproductive system and breast disorders) | 2 | 0
Fitz-hugh-curtis syndrome (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 — This SAE was assessed the investigators as related to study vaccination for one subject in the Havrix Group.
Hypertension (Vascular disorders) | 0 | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2 — This SAE was assessed the investigators as related to study vaccination for one subject in the Havrix Group.
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Malaria (Infections and infestations) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2
Tonsillitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 — This SAE was assessed the investigators as related to study vaccination for one subject in the Herpes Simplex Virus Group.
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 — This SAE was assessed the investigators as related to study vaccination for one subject in the Havrix Group.
Anxiety (Psychiatric disorders) | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 1
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Bipolar ii disorder (Psychiatric disorders) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1
Chlamydial cervicitis (Infections and infestations) | 0 | 1
Chorioamnionitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Complicated migraine (Nervous system disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Corneal abscess (Infections and infestations) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Death neonatal (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 1 | 0 — This SAE was assessed the investigators as related to study vaccination for one subject in the Herpes Simplex Virus Group.
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypothyroidic goitre (Endocrine disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Neurofibrosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ophthalmoplegic migraine (Nervous system disorders) | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Prophylaxis against hiv infection (Surgical and medical procedures) | 0 | 1
Removal of foreign body (Surgical and medical procedures) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 — This SAE was assessed the investigators as related to study vaccination for one subject in the Havrix Group.
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Stupor (Nervous system disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0 — This SAE was fatal and assessed by the investigators as not related to study vaccination.
Syncope (Nervous system disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 — This SAE was assessed the investigators as related to study vaccination for one subject in the Herpes Simplex Virus Group.
Tachycardia (Cardiac disorders) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tick-borne fever (Infections and infestations) | 1 | 0
Toxic shock syndrome (Infections and infestations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Ureteral polyp (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vaginal abscess (Infections and infestations) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Water intoxication (Metabolism and nutrition disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Herpes Simplex Virus Group (N=4488) | Havrix Group (N=3662)
Pain (General disorders) | 3902 | 2559
Redness (General disorders) | 1621 | 702
Swelling (General disorders) | 1371 | 438
Fatigue (General disorders) | 2031 | 1503
Headache (General disorders) | 1885 | 1456
Malaise (General disorders) | 1459 | 1003
Fever (General disorders) | 400 | 260
Upper respiratory tract infection (Infections and infestations) | 2154 | 1677

LIMITATIONS AND CAVEATS:
Out of the 8323 subjects enrolled and vaccinated, 7850 subjects were followed throughout the study, e. a. for safety and adverse event assessment (4488 in the Herpes Simplex Virus Group and 3662 in the Havrix Group).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.